CLINICAL TRIAL: NCT02923115
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled, Multi-Center, Single Ascending Dose Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of DS-1040b When Added to Standard of Care Anticoagulation Therapy in Subjects With Acute Submassive Pulmonary Embolism
Brief Title: Study to Assess the Safety, Pharmacokinetics/Dynamics of DS-1040b in Subjects With Acute Submassive Pulmonary Embolism
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DS1040-B-U107; 2015-005211-32 (EudraCT Number)
Record Dates: First submitted 2016-09-30; First posted 2016-10-04 (Estimated); Results first posted 2020-07-30 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Pulmonary Embolism; Thrombotic Disease
Keywords: Venous thromboembolism (VTE); Pulmonary embolism (PE); Acute Submassive Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism; Venous Thromboembolism | interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DS-1040b (Experimental): Participants who are randomized to receive DS-1040b as a single, continuous intravenous infusion (initial loading dose 3-6 mg). All participants will also receive standard of care anticoagulation enoxaparin therapy during the study drug infusion.
  Interventions: Drug: DS-1040b; Drug: Enoxaparin
- Placebo (Placebo Comparator): Participants who are randomized to receive placebo as a single, continuous intravenous infusion. All participants will also receive standard of care anticoagulation enoxaparin therapy during the study drug infusion.
  Interventions: Drug: Placebo; Drug: Enoxaparin

INTERVENTIONS:
Drug: DS-1040b — Single, continuous intravenous infusion over 12 to 24 hours (depending on cohort)
  Arms: DS-1040b
Drug: Placebo — Single, continuous intravenous infusion of 0.9% sodium chloride over 12 to 24 hours
  Arms: Placebo
Drug: Enoxaparin — Subcutaneous injection 1 mg/kg twice daily

SUMMARY:
This is a Phase 1b, double-blind (participants and Investigators), placebo-controlled, randomized, single-ascending dose, multi-center study to assess the safety, efficacy, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of DS-1040b in participants with acute submassive pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, age 18 to 75 years admitted to hospital with a clinical diagnosis of acute pulmonary embolism (PE) categorized as low risk or intermediate-risk or submassive PE and for whom catheter-based therapy is not planned;
* Subjects must have a computed tomography angiography (CTA) scan confirming the PE diagnosis and with at least one measurable index lesion in a segmental or larger pulmonary artery prior to randomization;
* Subjects should be in otherwise satisfactory health in the opinion of the Investigator;
* Subjects must be able to provide written informed consent.

Exclusion Criteria:

* Subjects with acute PE categorized as high-risk or massive, or who are hemodynamically unstable, evidenced by a heart rate > 120 /min and a systolic blood pressure (SBP) of < 90 mmHg for more than 15 consecutive minutes or a drop in SBP of > 40 mmHg since presentation;
* Subjects for whom use of a thrombolytic, either systemic or via catheter, is planned;
* Subjects with PE lesions only in the sub-segmental or smaller arteries;
* Subjects receiving any vitamin K antagonists (VKAs) prior to randomization or receiving more than 36 hours treatment with low molecular weight (LMW) Heparin in therapeutic doses prior to randomization;
* Subjects who had a prior intracranial hemorrhage, known arteriovenous malformation or aneurysm, head trauma, or evidence of active bleeding;
* Subjects who within 48 hours of randomization have used an anti-Factor IIa agent such as dabigatran or an anti-FXa agent such as rivaroxaban, apixaban, or edoxaban;
* Subjects who within 21 days prior to randomization have had gastrointestinal or genitourinary bleeding;
* Subjects who within 14 days prior to randomization have had major surgery or a lumbar puncture (or epidural steroid injection);
* Subjects with diagnosed active liver disease or with elevation of liver enzymes/bilirubin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (46):
- United States (15):
  - Pulmonary Associates of Mobile, Mobile, Alabama
  - Cedars-Sinai Medical Center, Beverly Hills, California
  - University of California, San Diego (UCSD) Medical Center, San Diego, California
  - Intercoastal Medical Group, Sarasota, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Mercury Street Medical, Butte, Montana
  - NYU Radiology Associate, New York, New York
  - Jacobi Medical Center, The Bronx, New York
  - Duke University Medical Center (DUMC), Durham, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Capital Area Research, Camp Hill, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
- Austria (3):
  - Medical University Graz, Graz
  - Medical University Innsbruck, Innsbruck
  - Medical University of Vienna, Vienna
- Belgium (3):
  - Universite Libre de Bruxelles (ULB) - Hopital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - University Hospital Leuven, Leuven
- France (6):
  - CHU de Brest - Hopital de la Cavale Blanche, Brest
  - CHU Gabriel Montpied Clermont-Ferrand, Clermont-Ferrand
  - CHU de Grenoble, La Tronche
  - Hopital Europeen Georges Pompidou, Paris
  - CHU St Etienne - Hopital Nord, Saint-Etienne
  - Hopital Civil de Strasbourg, Strasbourg
- Germany (5):
  - Staedtisches Klinikum Dresden-Friedrichstadt, Dresden
  - Universitaetsklinikum Dresden, Dresden
  - Universitaetsmedizin Greifswald, Greifswald
  - Universitatsklinikum Magdeburg, Magdeburg
  - Klinikum rechts der Isar, Technische Universität München, München
- Italy (4):
  - AOU Ospedali Riuniti di Ancona, Ancona
  - Universit degli Studi di Perugia - Azienda Ospedaliera di Perugia, Perugia
  - Humanitas Research Hospital, Rozzano
  - Ospedale di Circolo, Varese
- Netherlands (6):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Academisch Medisch Centrum, Amsterdam
  - Albert Schweitzer Hospital, Dordrecht
  - Leiden University Medical Center - Leids Universitair Medisch Centrum (LUMC), Leiden
  - HagaZiekenhuis, The Hague
  - UMC Utrecht, Utrecht
- Spain (4):
  - Hospital Universitario, Girona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 134 participants who met all inclusion and no exclusion criteria were enrolled in the study at 47 clinic sites (15 in the United States and 32 in Europe). Of the 134 participants randomized to treatment, 125 received treatment.
Pre-assignment Details: This study enrolled up to 5 sequential, ascending-dose, continuous infusion cohorts (starting DS1040b dose 20 mg). In Cohorts 1 and 2, eligible participants were randomized in a 2:1 ratio to either DS-1040b or placebo. Starting with Cohort 3, the ratio changed to 3:1. All participants received standard of care enoxaparin during study drug infusion.
Groups:
- Cohort 1: DS-1040b 20 mg: Participants who received an intravenous infusion of 20 mg DS-1040b in addition to standard of care anticoagulation therapy.
- Cohort 2: DS-1040b 40 mg; Cohort 5: DS-1040b 40 mg: Participants who received an intravenous infusion of 40 mg DS-1040b in addition to standard of care anticoagulation therapy.
- Cohort 3: DS-1040b 60 mg: Participants who received an intravenous infusion of 60 mg DS-1040b in addition to standard of care anticoagulation therapy.
- Cohort 4: DS-1040b 80 mg: Participants who received an intravenous infusion of 80 mg DS-1040b in addition to standard of care anticoagulation therapy.
- Placebo: Participants who received an intravenous infusion of placebo in addition to standard of care anticoagulation therapy.
Period: Overall Study
Arm/Group | Cohort 1: DS-1040b 20 mg | Cohort 2: DS-1040b 40 mg | Cohort 3: DS-1040b 60 mg | Cohort 4: DS-1040b 80 mg | Cohort 5: DS-1040b 40 mg | Placebo
Started (Randomized) | 12 | 16 | 23 | 23 | 22 | 38
Treated | 12 | 16 | 20 | 22 | 17 | 38
Completed | 12 | 15 | 20 | 21 | 17 | 38
Not Completed | 0 | 1 | 3 | 2 | 5 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Randomized, but not dosed | 0 | 0 | 3 | 1 | 5 | 0

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were assessed in the Safety Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: DS-1040b 20 mg | Cohort 2: DS-1040b 40 mg | Cohort 3: DS-1040b 60 mg | Cohort 4: DS-1040b 80 mg | Cohort 5: DS-1040b 40 mg | Placebo | Total
Number analyzed (Participants) | 12 | 16 | 20 | 22 | 17 | 38 | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 12 | 15 | 14 | 23 | 79
  >=65 years | 4 | 9 | 8 | 7 | 3 | 15 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (16.3) | 62.1 (10.9) | 55.1 (17.5) | 55.0 (13.5) | 56.5 (9.8) | 58.3 (10.7) | 57.2 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 4 | 7 | 5 | 12 | 40
  Male | 8 | 8 | 16 | 15 | 12 | 26 | 85
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1 | 3 | 5
  White | 12 | 15 | 19 | 22 | 16 | 34 | 118
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adjudicated Clinically Relevant Bleeding Events Following Intravenous Infusion of DS-1040b or Placebo in Addition to Standard of Care Anti-coagulation Therapy in Participants With Acute Submassive Pulmonary Embolism
Description: Clinically relevant bleeding was defined as major or clinically relevant non-major (CRNM) bleeding adjudicated by the Clinical Events Committee (CEC) based on International Society of Thrombosis and Haemostasis (ISTH) definitions and the CEC charter.
Time Frame: Baseline up to Day 30 post infusion, up to approximately 3 years 2 months
Population: Adjudicated bleeding events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: DS-1040b 20 mg | Cohort 2: DS-1040b 40 mg | Cohort 3: DS-1040b 60 mg | Cohort 4: DS-1040b 80 mg | Cohort 5: DS-1040b 40 mg | Placebo
Number analyzed (Participants) | 12 | 16 | 20 | 22 | 17 | 38
Participants
  At least 1 bleeding event | 4 | 3 | 3 | 4 | 1 | 10
  Major bleeding event | 0 | 0 | 0 | 1 | 0 | 0
  Non-major clinically relevant bleeding event | 0 | 0 | 0 | 2 | 1 | 1
  Minor or nuisance bleeding event | 3 | 2 | 3 | 2 | 0 | 6
  Fatal bleeding event | 0 | 0 | 0 | 0 | 0 | 0
  Bleeding with Hb drop ≥2g/dL, transfusion ≥2 units | 0 | 0 | 0 | 1 | 0 | 0

2. Secondary Outcome: Mean Percent Change From Baseline in Total Thrombus Volume at 12-72 Hours Post Start of Infusion of DS-1040b Compared to Placebo When Added to Standard of Care Anticoagulation Therapy in Participants With Acute Submassive Pulmonary Embolism
Description: The change from baseline in total thrombus volume was assessed by computed tomography angiography in segmental or larger pulmonary arteries following intravenous infusion of DS-1040b or placebo in addition to standard of care anti-coagulation therapy.
Time Frame: Baseline to 12-72 hours post start of infusion, up to approximately 3 years 2 months
Population: Changes in total thrombus volume were assessed in the Efficacy Analysis Set.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1: DS-1040b 20 mg | Cohort 2: DS-1040b 40 mg | Cohort 3: DS-1040b 60 mg | Cohort 4: DS-1040b 80 mg | Cohort 5: DS-1040b 40 mg | Placebo
Number analyzed (Participants) | 11 | 15 | 20 | 22 | 16 | 36
percent change | -23.78 (24.49) | -38.67 (17.34) | -33.50 (17.41) | -37.36 (26.90) | -32.33 (19.03) | -31.35 (17.74)

3. Secondary Outcome: Participants Achieving Reductions in Total Thrombus Volume at 12-72 Hours Post Infusion of DS-1040b Compared to Placebo When Added to Standard of Care Anticoagulation Therapy in Participants With Acute Submassive Pulmonary Embolism
Description: Change in total pulmonary thrombus burden (total thrombus volume) was assessed by computed tomography pulmonary angiography (CTPA). All CTPA scans were evaluated by a central imaging laboratory in a blinded manner by radiologists.
Time Frame: Baseline to 12-72 hours post start of infusion, up to approximately 3 years 2 months
Population: Reductions in total thrombus volume were assessed in the Efficacy Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: DS-1040b 20 mg | Cohort 2: DS-1040b 40 mg | Cohort 3: DS-1040b 60 mg | Cohort 4: DS-1040b 80 mg | Cohort 5: DS-1040b 40 mg | Placebo
Number analyzed (Participants) | 12 | 15 | 20 | 22 | 17 | 38
Participants
  No change or increase | 2 | 0 | 1 | 0 | 1 | 3
  <20% reduction | 2 | 3 | 3 | 5 | 3 | 5
  ≥20% reduction | 7 | 12 | 16 | 17 | 12 | 28
  Missing data | 1 | 0 | 0 | 0 | 1 | 2

4. Secondary Outcome: Pharmacokinetic (PK) Parameter Maximum Concentration (CMax) Following Intravenous Infusion of DS-1040b in Addition to Standard of Care Anti-coagulation Therapy in Participants With Acute Submassive Pulmonary Embolism
Description: Plasma concentrations at each time point and PK parameter Cmax of DS 1040b was calculated using non-compartmental analysis.
Time Frame: Cohort 1: 0 up to 72 h post infusion; Cohorts 2 and 3: 0 up to 96 h post infusion; Cohort 4 and 5: 0 up to 120 h post infusion
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: DS-1040b 20 mg | Cohort 2: DS-1040b 40 mg | Cohort 3: DS-1040b 60 mg | Cohort 4: DS-1040b 80 mg | Cohort 5: DS-1040b 40 mg
Number analyzed (Participants) | 11 | 15 | 19 | 22 | 17
ng/mL | 970.09 (1373.43) | 421.73 (515.57) | 608.84 (562.94) | 1006.41 (1883.49) | 526.12 (535.03)

5. Secondary Outcome: Pharmacokinetic Parameter Area Under the Concentration Versus Time Curve (0 to Last) Following Intravenous Infusion of DS-1040b In Addition to Standard of Care Anti-coagulation Therapy in Participants With Acute Submassive Pulmonary Embolism
Description: Plasma concentrations at each time point and PK parameter of Area Under the Concentration Versus Time Curve (0 to last) of DS-1040b was calculated using non-compartmental analysis.
Time Frame: as for outcome 4
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort 1: DS-1040b 20 mg | Cohort 2: DS-1040b 40 mg | Cohort 3: DS-1040b 60 mg | Cohort 4: DS-1040b 80 mg | Cohort 5: DS-1040b 40 mg
Number analyzed (Participants) | 11 | 15 | 19 | 22 | 17
ng*h/mL | 5532.92 (4090.34) | 7819.53 (2870.13) | 13403.15 (8047.13) | 17147.27 (15024.61) | 8014.73 (2870.19)

6. Secondary Outcome: Pharmacokinetic Parameter Terminal Half-life Following Intravenous Infusion of DS-1040b Combined With Standard of Care Anti-coagulation Therapy in Participants With Acute Submassive Pulmonary Embolism
Description: Plasma concentrations at each time point and PK parameter Terminal Half-life of DS-1040b was calculated using non-compartmental analysis.
Time Frame: as for outcome 4
Population: Terminal half-life was assessed in patients with available data in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1: DS-1040b 20 mg | Cohort 2: DS-1040b 40 mg | Cohort 3: DS-1040b 60 mg | Cohort 4: DS-1040b 80 mg | Cohort 5: DS-1040b 40 mg
Number analyzed (Participants) | 9 | 13 | 18 | 5 | 9
hours | 22.81 (3.13) | 28.44 (5.75) | 29.06 (7.60) | 36.39 (2.07) | 30.06 (3.45)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from baseline up to Day 30 post infusion, up to approximately 3 years 2 months.
Description: A TEAE is defined as an adverse event that emerges during treatment, having been absent pretreatment, or worsening relative to the pre-treatment state.
Arm/Group | Cohort 1: DS-1040b 20 mg | Cohort 2: DS-1040b 40 mg | Cohort 3: DS-1040b 60 mg | Cohort 4: DS-1040b 80 mg | Cohort 5: DS-1040b 40 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/16 | 0/20 | 0/22 | 0/17 | 0/38
Serious Adverse Events (participants affected / at risk) | 3/12 | 0/16 | 2/20 | 1/22 | 3/17 | 5/38
Other Adverse Events (participants affected / at risk) | 8/12 | 6/16 | 13/20 | 10/22 | 8/17 | 25/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: DS-1040b 20 mg (N=12) | Cohort 2: DS-1040b 40 mg (N=16) | Cohort 3: DS-1040b 60 mg (N=20) | Cohort 4: DS-1040b 80 mg (N=22) | Cohort 5: DS-1040b 40 mg (N=17) | Placebo (N=38)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Metastases to nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Testicular cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: DS-1040b 20 mg (N=12) | Cohort 2: DS-1040b 40 mg (N=16) | Cohort 3: DS-1040b 60 mg (N=20) | Cohort 4: DS-1040b 80 mg (N=22) | Cohort 5: DS-1040b 40 mg (N=17) | Placebo (N=38)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 0 | 0 | 3
Headache (Nervous system disorders) | 1 | 0 | 3 | 2 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 1 | 2
Lung infection (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Metastases to nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Testicular cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 1 | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Infusion site phlebitis (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Liver function test increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasticity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Right ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ketonuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Crystal urine present (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram ST segment abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Mean cell volume increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Occult blood positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Urobilinogen urine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Sinus operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-21): https://cdn.clinicaltrials.gov/large-docs/15/NCT02923115/Prot_SAP_000.pdf